CLINICAL TRIAL: NCT04712604
Title: Feasibility and Acceptability Study of My Sleep Our Sleep (MSOS) Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Youngmee Kim, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20201067
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Insomnia
Keywords: Sleep disturbance in GI cancer patients and their sleep partner
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSOS Group (Experimental): The participants in this group will receive the MSOS Intervention for 4 consecutive weeks.
  Interventions: Behavioral: My Sleep Our Sleep (MSOS) Program

INTERVENTIONS:
Behavioral: My Sleep Our Sleep (MSOS) Program — MSOS Program is a weekly one-hour Zoom session that focuses on psychoeducation on sleep health for both patients and their sleep partners.

SUMMARY:
The purpose of this study is to test feasibility and acceptability of a psycho-behavioral intervention on sleep in cancer patients and their partners.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. newly diagnosed with a gastrointestinal cancer (stage I to IV) 12 months or less prior to participating
2. 18 years or older
3. able to speak/read English at the 5th grade level
4. having a consistent partner who is involved in daily activities including sleep
5. having 5 or greater score on the Pittsburgh Sleep Quality Index.

Sleep partners:

1. 18 years or older
2. able to speak/read English at the 5th grade level
3. a partner of the patient who is involved in the patient's daily activities including sleep
4. having similar circadian rhythm/sleep patterns with the patient
5. having 5 or greater score on the Pittsburgh Sleep Quality Index.

Exclusion Criteria:

Patients and their sleep partners:

1. having had a diagnosis of dementia, psychotic disorder, major depressive disorder, bipolar disorder, which currently has not been treated
2. having active suicidality in the past year
3. currently having an untreated diagnosed sleep disorder (narcolepsy, restless leg syndrome)
4. currently having have a poor physical functioning status as measured by an Eastern Cooperative Oncology Group (ECOG) score of 3 or higher and Karnofsky grade of 50 or lower
5. having poor cognitive function status as measured by the Mini Mental State Examination score of 24 or less
6. unable to see or hear
7. at the end of life (life expectancy of less than a month)
8. unwilling to change their current sleep-related habits in near future.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-03-14 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Feasibility of the intervention | 4 weeks
  Feasibility of the intervention will be reported as the percentage of participants who enroll and complete all the sessions of the study.
Acceptability of the intervention | 4 weeks
  Acceptability of the intervention will be reported as the percentage of participants who evaluated the intervention and the interventionist as "satisfactory" or better.

SECONDARY OUTCOMES:
Change in sleep disturbance | Baseline, 4 weeks
  Change in sleep disturbance as measured by the Pittsburgh Sleep Quality Index (PSQI). PSQI has a total score ranging from 0 to 21, where lower score indicates healthier sleep quality.
Change in quality of life | Baseline, 4 weeks
  Change in quality of life as measured by the Patient-reported Outcomes Measurement Information System (PROMIS-29). PROMIS-29 has a total score ranging from 20-80, with lower scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Youngmee Kim, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim Y, Ting A, Tsai TC, Carver CS. Dyadic sleep intervention for adult patients with cancer and their sleep-partner caregivers: A feasibility study. Palliat Support Care. 2024 Apr;22(2):226-235. doi: 10.1017/S1478951523000627. PMID 37312582
- [Derived] Kim Y, Ting A, Steel JL, Tsai TC. Protocol of a dyadic sleep intervention for adult patients with cancer and their sleep-partner caregivers. Contemp Clin Trials Commun. 2023 Jan 16;32:101064. doi: 10.1016/j.conctc.2023.101064. eCollection 2023 Apr. PMID 36704757